CLINICAL TRIAL: NCT01385969
Title: Using the Natural Recoil of the Inflating Syringe as a Safety Valve to Limit LMA Cuff Pressure and Decrease LMA-Induced Complications
Brief Title: LMA Cuff Pressure and LMA-induced Complications
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christopher B. Robards, MD, Mayo Clinic
Other Study IDs: 11-001506
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Sore Throat; Dysphagia; Dysphonia
Keywords: overinflation of LMAs
MeSH Terms: conditions — Pharyngitis; Deglutition Disorders; Dysphonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Standard Practice
  Interventions: Device: Standard inflation of LMA cuff
- Syringe recoil
  Interventions: Device: Pressure check with syringe recoil
- Pressure Transducer
  Interventions: Device: Pressure check by pressure transducer

INTERVENTIONS:
Device: Standard inflation of LMA cuff — LMA cuff will be inflated per standard practice with a syringe and resulting cuff pressure will be measured by manual palpation of the cuff per standard practice.
  Other Names: LMA inflation routine clinical practice
  Groups: Standard Practice
Device: Pressure check with syringe recoil — LMA cuff will be inflated per standard practice with a syringe and resulting cuff pressure will be measured by syringe recoil
  Other Names: LMA cuff pressure by syringe recoil
  Groups: Syringe recoil
Device: Pressure check by pressure transducer — LMA cuff will be inflated per standard practice with a syringe and resulting cuff pressure will be measured by pressure transducer.
  Other Names: LMA cuff pressure checked by pressure transducer
  Groups: Pressure Transducer

SUMMARY:
The purpose of this study is to determine if using 20 mL B.Braun syringes to inflate LMAs and allowing them to recoil will put the pressure of the LMA cuff within the safety range. It will also determine if remaining within this safety range has an effect on complications after surgery..

ELIGIBILITY:
Inclusion Criteria:

* Registered Mayo Clinic in Florida patients scheduled to undergo a surgery
* Planned use of LMA during surgery
* between the ages of 18-99
* short duration (<2 hours elective surgery)

Exclusion Criteria:

* recent history of upper respiratory tract infection
* intra-cavitary or laparoscopic procedure
* risk of pulmonary aspiration
* known difficult airway
* history of gastric reflux
* BMI > 40
* lateral or prone positions
* oral or nasal surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo a surgical procedure less than 2 hours in duration
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2011-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pressure of the syringe after inflation of the LMA cuff | after inflation, 1 hour into surgery

SECONDARY OUTCOMES:
Number of patients with dysphagia and/or dysphonia | 1, 2, and 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Robards, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - University of Florida College of Medicine, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida